CLINICAL TRIAL: NCT05955430
Title: Efficacy of Percutaneous Electrical Stimulation Compared to Transcutaneous Electrical Stimulation in Combination With an Education and Exercise Program in Patients With Knee Osteoarthritis
Brief Title: Percutaneous Electrical Stimulation, Education and Exercise Program in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Josue Fernandez Carnero (Other)
Responsible Party: Sponsor-Investigator, Josue Fernandez Carnero, Professor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KOA1
Record Dates: First submitted 2023-07-05; First posted 2023-07-21 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Physiotherapy; Physical Therapy; Conditioned Pain Modulation; Temporal Summation of pain; Knee pain; PENS; Percutaneous electrical stimulation; Pain education
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise, education and PENS (Experimental): Patients will receive eight face-to-face sessions of therapeutic exercise, four sessions of pain education and eight sessions of percutaneous electrical stimulation (PENS).
  Interventions: Other: Therapeutic exercise; Other: Pain education; Other: Percutaneous electrical stimulation
- Exercise, education and TENS (Active Comparator): Patients will receive eight face-to-face sessions of therapeutic exercise, four sessions of pain education and eight sessions of transcutaneous electrical stimulation (TENS).
  Interventions: Other: Therapeutic exercise; Other: Pain education; Other: Transcutaneous electrical stimulation
- Exercise, education and placebo stimulation (Placebo Comparator): Patients will receive eight face-to-face sessions of therapeutic exercise, four sessions of pain education and eight sessions of placebo stimulation.
  Interventions: Other: Therapeutic exercise; Other: Pain education; Other: Placebo stimulation

INTERVENTIONS:
Other: Therapeutic exercise — It consists of strengthening exercises and gradual walking. The lower limb strengthening exercises are individualized and progressive for each patient for twelve weeks. There will be eight face-to-face sessions over four weeks. And then the patient will continue with those exercises for eight more weeks. In addition, they must perform twelve weeks of progressive walking until they are walking at least 30 minutes, 5 days a week at a moderate intensity (defined as moderate shortness of breath while walking).
Other: Pain education — A therapeutic pain education program for patients will be implemented. There will be four 30-minute face-to-face sessions (one session per week). The objective is to change the participants' conceptualization of pain. From seeing pain as a marker of tissue damage to a marker of the body's perceived need for protection. Contents include basic structure of the nervous system, distinction between nociception and pain, peripheral and central sensitization, neuroplasticity and benefits of exercise.
Other: Percutaneous electrical stimulation — A TENS (100 Hz 100 ms) current will be applied through four needles located in the knee for 30 minutes. Eight sessions will be held during a month (two per week). The distribution of the channels will be for the first channel anode in lateral anterior zone and cathode in medial anterior zone and for the second channel anode in Hoffa's fat and cathode in goose foot. Participants will be able to adjust the amplitude to a strong and manageable sensory stimulation intensity that was not strong enough to cause muscle contraction.
  Arms: Exercise, education and PENS
Other: Transcutaneous electrical stimulation — A TENS (100 Hz 100 ms) current will be applied through four patches located in the knee for 30 minutes. Eight sessions will be held during a month (two per week). The distribution of the channels will be for the first channel anode in lateral anterior zone and cathode in medial anterior zone and for the second channel anode in Hoffa's fat and cathode in goose foot. Participants will be able to adjust the amplitude to a strong and manageable sensory stimulation intensity that was not strong enough to cause muscle contraction.
  Arms: Exercise, education and TENS
Other: Placebo stimulation — To perform the dry needling placebo, modified needles will be used according to the validation performed by Mitchell et al. 2018, since they generate more puncture sensation than normal needles, which has been shown to generate more analgesia and to be more effective as a placebo. To perform placebo TENS, the protocol established by Rakel et al. 2010 will be used, which consists of applying a TENS of 100 Hz and 100 ms for 30 seconds and then lowering the intensity during the following 15 seconds. Eight sessions will be held during a month (two per week).
  Arms: Exercise, education and placebo stimulation

SUMMARY:
The purpose of this study is to compare the effectiveness of percutaneous electrotherapy treatment with transcutaneous and placebo.

DETAILED DESCRIPTION:
There is evidence of the benefit of therapeutic exercise on pain intensity and functionality in patients with osteoarthritis of the knee. However, there is a lack of evidence of its effectiveness when applied in combination with new treatment strategies such as percutaneous electrostimulation and therapeutic pain education.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 45 years
* Have activity related joint pain
* Have morning stiffness ≤30 min
* Knee pain of at least 6 months duration
* OA diagnosis by physician
* Current levels of moderate/vigorous physical activity (MVPA) below physical activity guideline recommendations (< 150 min/week of MVPA; assessed using the Active Australia Physical Activity Questionnaire)

Exclusion Criteria:

* Health conditions that prevent safe participation in physical activity interventions as listed in the American College of Sports Medicine Guidelines (e.g., cardiac or lung disease).
* Pain in other body areas that currently limits walking ability (e.g., back pain, foot pain, hip pain)
* Neurological disorders affecting lower limb movement (e.g., multiple sclerosis or stroke).
* Inflammatory arthritis (including rheumatoid arthritis)
* Fibromyalgia
* Previously operated knee is the most painful knee
* Any condition impacting decision-making/memory (e.g., Alzheimer's, dementia)
* Severe depression
* Current moderate/vigorous physical activity levels above guideline recommendations (≥150 min/week; assessed using the Active Australia Physical Activity Questionnaire)
* Currently undergoing regular, active intervention for the knee (e.g., seeing a physiotherapist)
* Unable to commit to study requirements (unable to attend study appointments or complete study outcomes)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to one month in WOMAC | At baseline and at one month
  The Western Ontario and McMaster (WOMAC) Universities Osteoarthritis Index is a specific questionnaire for knee and hip osteoarthritis that assesses pain, stiffness and functional capacity, currently recommended by several international organizations for the evaluation of this disease.
Change from baseline to three months in WOMAC | At baseline and at three months
  The Western Ontario and McMaster (WOMAC) Universities Osteoarthritis Index is a specific questionnaire for knee and hip osteoarthritis that assesses pain, stiffness and functional capacity, currently recommended by several international organizations for the evaluation of this disease.
Change from baseline to six months in WOMAC | At baseline and at six months
  The Western Ontario and McMaster (WOMAC) Universities Osteoarthritis Index is a specific questionnaire for knee and hip osteoarthritis that assesses pain, stiffness and functional capacity, currently recommended by several international organizations for the evaluation of this disease.
Change from baseline to immediately after the first session in VAS | At baseline and immediately after the first session
  The visual analogue scale (VAS) uses a 10 cm line with endpoint descriptors such as 'no pain' marked at the left end of the line and 'worst pain imaginable' marked at the right end. Patients are asked to mark a point on the line that best represents their pain.
Change from baseline to one month in VAS | At baseline and at one month
  The visual analogue scale (VAS) uses a 10 cm line with endpoint descriptors such as 'no pain' marked at the left end of the line and 'worst pain imaginable' marked at the right end. Patients are asked to mark a point on the line that best represents their pain.
Change from baseline to three months in VAS | At baseline and at three months
  The visual analogue scale (VAS) uses a 10 cm line with endpoint descriptors such as 'no pain' marked at the left end of the line and 'worst pain imaginable' marked at the right end. Patients are asked to mark a point on the line that best represents their pain.
Change from baseline to six months in VAS | At baseline and at six months
  The visual analogue scale (VAS) uses a 10 cm line with endpoint descriptors such as 'no pain' marked at the left end of the line and 'worst pain imaginable' marked at the right end. Patients are asked to mark a point on the line that best represents their pain.

SECONDARY OUTCOMES:
Change from baseline to immediately after the first session in PPT | At baseline and immediately after the first session
  Pressure Pain Threshold (PPT) will be assessed at thumb, trapezius superior muscle, tibialis anterior muscle and patella using a digital algometer (Wagner instruments, Greenwich, CT, USA). Participants will be instructed to say "stop" when the pressure sensation becomes painful. The average of two trials for each side will be performed for analysis. The algometer pressure for assessment will be gradually increased at a rate of 1kg/second. Data will be collected in kg/cm2.
Change from baseline to one month in PPT | At baseline and at one month
  Pressure Pain Threshold (PPT) will be assessed at thumb, trapezius superior muscle, tibialis anterior muscle and patella using a digital algometer (Wagner instruments, Greenwich, CT, USA). Participants will be instructed to say "stop" when the pressure sensation becomes painful. The average of two trials for each side will be performed for analysis. The algometer pressure for assessment will be gradually increased at a rate of 1kg/second. Data will be collected in kg/cm2.
Change from baseline to three months in PPT | At baseline and at three months
  Pressure Pain Threshold (PPT) will be assessed at thumb, trapezius superior muscle, tibialis anterior muscle and patella using a digital algometer (Wagner instruments, Greenwich, CT, USA). Participants will be instructed to say "stop" when the pressure sensation becomes painful. The average of two trials for each side will be performed for analysis. The algometer pressure for assessment will be gradually increased at a rate of 1kg/second. Data will be collected in kg/cm2.
Change from baseline to six months in PPT | At baseline and at six months
  Pressure Pain Threshold (PPT) will be assessed at thumb, trapezius superior muscle, tibialis anterior muscle and patella using a digital algometer (Wagner instruments, Greenwich, CT, USA). Participants will be instructed to say "stop" when the pressure sensation becomes painful. The average of two trials for each side will be performed for analysis. The algometer pressure for assessment will be gradually increased at a rate of 1kg/second. Data will be collected in kg/cm2.
Change from baseline to immediately after the first session in CPM | At baseline and immediately after the first session
  Conditioned pain modulation (CPM) is a centrally processed measure of the net effect of the descending pain pathway. A digital algometer will be used for the test stimulus and a pressure cuff will be used for the conditioned stimulus. Pain intensity will be measured with the numeric rating scale (NRS).
Change from baseline to one month in CPM | At baseline and at one month
  Conditioned pain modulation (CPM) is a centrally processed measure of the net effect of the descending pain pathway. A digital algometer will be used for the test stimulus and a pressure cuff will be used for the conditioned stimulus. Pain intensity will be measured with the numeric rating scale (NRS).
Change from baseline to three months in CPM | At baseline and at three months
  Conditioned pain modulation (CPM) is a centrally processed measure of the net effect of the descending pain pathway. A digital algometer will be used for the test stimulus and a pressure cuff will be used for the conditioned stimulus. Pain intensity will be measured with the numeric rating scale (NRS).
Change from baseline to six months in CPM | At baseline and at six months
  Conditioned pain modulation (CPM) is a centrally processed measure of the net effect of the descending pain pathway. A digital algometer will be used for the test stimulus and a pressure cuff will be used for the conditioned stimulus. Pain intensity will be measured with the numeric rating scale (NRS).
Change from baseline to immediately after the first session in TSP | At baseline and immediately after the first session
  Temporal summation of pain (TSP) is a noninvasive and indirect measure of central sensitization in humans, which refers to an increase in pain intensity with repetitive noxious stimuli. An Algometer will be used to induce temporal summation. It will be applied vertically, directly on the thumb on the asymptomatic side, stimulating 10 consecutive times for 1 second and with 1 second intervals with a previously determined pressure. The results will be obtained by the difference between the first and the tenth measurement of pain intensity.
Change from baseline to one month in TSP | At baseline and at one month
  Temporal summation of pain (TSP) is a noninvasive and indirect measure of central sensitization in humans, which refers to an increase in pain intensity with repetitive noxious stimuli. An Algometer will be used to induce temporal summation. It will be applied vertically, directly on the thumb on the asymptomatic side, stimulating 10 consecutive times for 1 second and with 1 second intervals with a previously determined pressure. The results will be obtained by the difference between the first and the tenth measurement of pain intensity.
Change from baseline to three months in TSP | At baseline and at three months
  Temporal summation of pain (TSP) is a noninvasive and indirect measure of central sensitization in humans, which refers to an increase in pain intensity with repetitive noxious stimuli. An Algometer will be used to induce temporal summation. It will be applied vertically, directly on the thumb on the asymptomatic side, stimulating 10 consecutive times for 1 second and with 1 second intervals with a previously determined pressure. The results will be obtained by the difference between the first and the tenth measurement of pain intensity.
Change from baseline to six months in TSP | At baseline and at six months
  Temporal summation of pain (TSP) is a noninvasive and indirect measure of central sensitization in humans, which refers to an increase in pain intensity with repetitive noxious stimuli. An Algometer will be used to induce temporal summation. It will be applied vertically, directly on the thumb on the asymptomatic side, stimulating 10 consecutive times for 1 second and with 1 second intervals with a previously determined pressure. The results will be obtained by the difference between the first and the tenth measurement of pain intensity.
Change from baseline to one month in TUG | At baseline and at one month
  The Timed Up and Go (TUG) Test is a test especially indicated to measure mobility and assess the risk of falls in the elderly. The patient will begin sitting in a chair with his back supported and his arms on the armrests, when he hears the word "Let's go" he must get up and walk to a mark that will be on the ground 3 meters away and finally the person will turn around and walk again to sit on the chair. The time it takes from when you say "Let's go" until he sits down again will be timed (3 attempts and the results are averaged).
Change from baseline to three months in TUG | At baseline and at three months
  The Timed Up and Go (TUG) Test is a test especially indicated to measure mobility and assess the risk of falls in the elderly. The patient will begin sitting in a chair with his back supported and his arms on the armrests, when he hears the word "Let's go" he must get up and walk to a mark that will be on the ground 3 meters away and finally the person will turn around and walk again to sit on the chair. The time it takes from when you say "Let's go" until he sits down again will be timed (3 attempts and the results are averaged).
Change from baseline to six months in TUG | At baseline and at six months
  The Timed Up and Go (TUG) Test is a test especially indicated to measure mobility and assess the risk of falls in the elderly. The patient will begin sitting in a chair with his back supported and his arms on the armrests, when he hears the word "Let's go" he must get up and walk to a mark that will be on the ground 3 meters away and finally the person will turn around and walk again to sit on the chair. The time it takes from when you say "Let's go" until he sits down again will be timed (3 attempts and the results are averaged).
Change from baseline to one month in GCPS | At baseline and at one month
  Pain severity will be assessed using the Spanish version of the Chronic Pain Grading Scale (GCPS). This scale is a self-reported instrument that consists of two subscales; the first assesses pain intensity, and the second assesses perceived disability. The scale is made up of a total of 8 items, 7 of which are 11 points in Likert format, and the other item assesses the perpetuation of pain, asking for the number of days of pain in the previous 6 months. The Spanish version of the GCPS has proven to be a valid and reliable instrument to assess the severity of chronic pain.
Change from baseline to three months in GCPS | At baseline and at three months
  Pain severity will be assessed using the Spanish version of the Chronic Pain Grading Scale (GCPS). This scale is a self-reported instrument that consists of two subscales; the first assesses pain intensity, and the second assesses perceived disability. The scale is made up of a total of 8 items, 7 of which are 11 points in Likert format, and the other item assesses the perpetuation of pain, asking for the number of days of pain in the previous 6 months. The Spanish version of the GCPS has proven to be a valid and reliable instrument to assess the severity of chronic pain.
Change from baseline to six months in GCPS | At baseline and at six months
  Pain severity will be assessed using the Spanish version of the Chronic Pain Grading Scale (GCPS). This scale is a self-reported instrument that consists of two subscales; the first assesses pain intensity, and the second assesses perceived disability. The scale is made up of a total of 8 items, 7 of which are 11 points in Likert format, and the other item assesses the perpetuation of pain, asking for the number of days of pain in the previous 6 months. The Spanish version of the GCPS has proven to be a valid and reliable instrument to assess the severity of chronic pain.
Baseline Mini-Mental Status | At baseline
  MEC is the spanish version of the Mini-Mental Status Examination. It is the most widely used cognitive screening test to assess suspected symptoms compatible with cognitive impairment or dementia. Through a series of questions and requests, different cognitive functions are evaluated: temporal and spatial orientation, immediate memory, information storage and retrieval, concentration and working memory, oral language, reading and writing a sentence and visoconstruction by copying a simple drawing.
Change from baseline to one month in STAI | At baseline and at one month
  The State-Trait Anxiety Inventory (STAI). This questionnaire comprises two subsections of 20 items each for the measurement of anxiety as a state and as a trait, with a 4-point Likert-type response (0: not at all; 3: very much). Scores range from 0 to 60 points, with higher scores indicating greater anxiety.
Change from baseline to three months in STAI | At baseline and at three months
  The State-Trait Anxiety Inventory (STAI). This questionnaire comprises two subsections of 20 items each for the measurement of anxiety as a state and as a trait, with a 4-point Likert-type response (0: not at all; 3: very much). Scores range from 0 to 60 points, with higher scores indicating greater anxiety.
Change from baseline to six months in STAI | At baseline and at six months
  The State-Trait Anxiety Inventory (STAI). This questionnaire comprises two subsections of 20 items each for the measurement of anxiety as a state and as a trait, with a 4-point Likert-type response (0: not at all; 3: very much). Scores range from 0 to 60 points, with higher scores indicating greater anxiety.
Change from baseline to one month in BDI-II | At baseline and at one month
  Beck Depression Inventory-II (BDI-II) is a self-report measure of depression in a variety of settings and populations. It is the most widely used questionnaire worldwide to assess depression. The total score ranges from 0 to 63 points. A change of 5 points corresponds to a minimally important clinical difference.
Change from baseline to three months in BDI-II | At baseline and at three months
  Beck Depression Inventory-II (BDI-II) is a self-report measure of depression in a variety of settings and populations. It is the most widely used questionnaire worldwide to assess depression. The total score ranges from 0 to 63 points. A change of 5 points corresponds to a minimally important clinical difference.
Change from baseline to six months in BDI-II | At baseline and at six months
  Beck Depression Inventory-II (BDI-II) is a self-report measure of depression in a variety of settings and populations. It is the most widely used questionnaire worldwide to assess depression. The total score ranges from 0 to 63 points. A change of 5 points corresponds to a minimally important clinical difference.
Change from baseline to one month in PCS | At baseline and at one month
  The Spanish version of the Pain Catastrophizing Scale (PCS) it has 13 items and each one is rated on a 5-point scale: 0 (not at all) to 4 (all the time). It comprises 3 dimensions: rumination, magnification, and despair. The theoretical range of the instrument is between 13 and 62, with low scores indicating low catastrophism and high values indicating high catastrophism.
Change from baseline to three months in PCS | At baseline and at three months
  The Spanish version of the Pain Catastrophizing Scale (PCS) it has 13 items and each one is rated on a 5-point scale: 0 (not at all) to 4 (all the time). It comprises 3 dimensions: rumination, magnification, and despair. The theoretical range of the instrument is between 13 and 62, with low scores indicating low catastrophism and high values indicating high catastrophism.
Change from baseline to six months in PCS | At baseline and at six months
  The Spanish version of the Pain Catastrophizing Scale (PCS) it has 13 items and each one is rated on a 5-point scale: 0 (not at all) to 4 (all the time). It comprises 3 dimensions: rumination, magnification, and despair. The theoretical range of the instrument is between 13 and 62, with low scores indicating low catastrophism and high values indicating high catastrophism.
Change from baseline to one month in TSK-11 | At baseline and at one month
  Tampa Scale for Kinesiophobia (TSK-11) is an 11-item scale that assesses the degree of fear of movement and (re)injury. Each item is scored from 1 to 4 according to the degree of agreement with the statement (1: do not agree at all; 4: strongly agree). The validated Spanish version of the 11-item scale has a total score of 11 to 44 items and has two subscales: activity avoidance and harm.
Change from baseline to three months in TSK-11 | At baseline and at three months
  Tampa Scale for Kinesiophobia (TSK-11) is an 11-item scale that assesses the degree of fear of movement and (re)injury. Each item is scored from 1 to 4 according to the degree of agreement with the statement (1: do not agree at all; 4: strongly agree). The validated Spanish version of the 11-item scale has a total score of 11 to 44 items and has two subscales: activity avoidance and harm.
Change from baseline to six months in TSK-11 | At baseline and at six months
  Tampa Scale for Kinesiophobia (TSK-11) is an 11-item scale that assesses the degree of fear of movement and (re)injury. Each item is scored from 1 to 4 according to the degree of agreement with the statement (1: do not agree at all; 4: strongly agree). The validated Spanish version of the 11-item scale has a total score of 11 to 44 items and has two subscales: activity avoidance and harm.
Change from baseline to immediately after the first intervention in catastrophism in vivo | At baseline and immediately after the first intervention
  In vivo catastrophism. Questions will be asked regarding the types of thoughts and feelings of the patient while the painful stimulus was applied in the measurement of conditioned pain modulation. Using the a scale, you are asked to indicate the degree to which you had these thoughts and feelings during the pain test.
Change from baseline to one month in CRES-4 | At baseline and at one month
  Consumer Reports Effectiveness Scale (CRES-4) consisting of four items designed to evaluate whether patients are satisfied with the therapy they have received and if it has been perceived as effective or not. Its global score is intended to reflect treatment effectiveness as perceived by the patient.
Change from baseline to three months in CRES-4 | At baseline and at three months
  Consumer Reports Effectiveness Scale (CRES-4) consisting of four items designed to evaluate whether patients are satisfied with the therapy they have received and if it has been perceived as effective or not. Its global score is intended to reflect treatment effectiveness as perceived by the patient.
Change from baseline to six months in CRES-4 | At baseline and at six months
  Consumer Reports Effectiveness Scale (CRES-4) consisting of four items designed to evaluate whether patients are satisfied with the therapy they have received and if it has been perceived as effective or not. Its global score is intended to reflect treatment effectiveness as perceived by the patient.
Change from baseline to one month in GROC | At baseline and at one month
  The Global Rating of Change Score (GRoC) is a frequently used outcome measure that has been used to independently score self-perceived improvement in a patient and has been used as an anchor method to determine minimal clinically important change scores. The GRoC is a single-item, recall-based questionnaire of well-being that is based on progress (or lack of progress) since an initial treatment encounter.
Change from baseline to three months in GROC | At baseline and at three months
  The Global Rating of Change Score (GRoC) is a frequently used outcome measure that has been used to independently score self-perceived improvement in a patient and has been used as an anchor method to determine minimal clinically important change scores. The GRoC is a single-item, recall-based questionnaire of well-being that is based on progress (or lack of progress) since an initial treatment encounter.
Change from baseline to six months in GROC | At baseline and at six months
  The Global Rating of Change Score (GRoC) is a frequently used outcome measure that has been used to independently score self-perceived improvement in a patient and has been used as an anchor method to determine minimal clinically important change scores. The GRoC is a single-item, recall-based questionnaire of well-being that is based on progress (or lack of progress) since an initial treatment encounter.
Baseline Demographic and Clinical Characteristics | At baseline
  Demographic information including sex, age, weight, height, pain duration, the mean and worse pain intensities during the last week using the Visual Analogue Scale will be collected.
Change from baseline to one month in SPPB | At baseline and at one month
  Short physical performance battery (SPPB). It makes it possible to classify the level of physical functioning of the elderly throughout the entire functional spectrum. It consists of carrying out three tests: balance (in three positions: feet together, semi-tandem and tandem), gait speed (4 meters) and getting up and sitting down on a chair five times.The total SPPB score and outcome assessment results from the sum of the three subtests, and ranges from 0 (worst) to 12; changes of 1 point have clinical significance. A score below 10 indicates frailty and an elevated risk of disability as well as falls.
Change from baseline to three months in SPPB | At baseline and at three months
  Short physical performance battery (SPPB). It makes it possible to classify the level of physical functioning of the elderly throughout the entire functional spectrum. It consists of carrying out three tests: balance (in three positions: feet together, semi-tandem and tandem), gait speed (4 meters) and getting up and sitting down on a chair five times. The total SPPB score and outcome assessment results from the sum of the three subtests, and ranges from 0 (worst) to 12; changes of 1 point have clinical significance. A score below 10 indicates frailty and an elevated risk of disability as well as falls.
Change from baseline to six months in SPPB | At baseline and at six months
  Short physical performance battery (SPPB). It makes it possible to classify the level of physical functioning of the elderly throughout the entire functional spectrum. It consists of carrying out three tests: balance (in three positions: feet together, semi-tandem and tandem), gait speed (4 meters) and getting up and sitting down on a chair five times. The total SPPB score and outcome assessment results from the sum of the three subtests, and ranges from 0 (worst) to 12; changes of 1 point have clinical significance. A score below 10 indicates frailty and an elevated risk of disability as well as falls.
Change from baseline to one month in SF-12 | At baseline and at one month
  The SF-12 Health Survey (SF-12) is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective. Generic patient-reported outcome measures like the SF-12 assess general health and well-being, including the impact of any and all illnesses on a broad range of functional domains. The response options form Likert-type scales (where the number of options varies from three to six points, depending on the item), which evaluate intensity and/or frequency of people's health status. The score ranges from 0 to 100, where the higher the score, the better the health-related quality of life.
Change from baseline to three months in SF-12 | At baseline and at three months
  The SF-12 Health Survey (SF-12) is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective. Generic patient-reported outcome measures like the SF-12 assess general health and well-being, including the impact of any and all illnesses on a broad range of functional domains. The response options form Likert-type scales (where the number of options varies from three to six points, depending on the item), which evaluate intensity and/or frequency of people's health status. The score ranges from 0 to 100, where the higher the score, the better the health-related quality of life.
Change from baseline to six months in SF-12 | At baseline and at six months
  The SF-12 Health Survey (SF-12) is a 12-item questionnaire used to assess generic health outcomes from the patient's perspective. Generic patient-reported outcome measures like the SF-12 assess general health and well-being, including the impact of any and all illnesses on a broad range of functional domains. The response options form Likert-type scales (where the number of options varies from three to six points, depending on the item), which evaluate intensity and/or frequency of people's health status. The score ranges from 0 to 100, where the higher the score, the better the health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Josué Fernández Carnero, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stanton TR, Braithwaite FA, Butler D, Moseley GL, Hill C, Milte R, Ratcliffe J, Maher C, Tomkins-Lane C, Pulling BW, MacIntyre E, Esterman A, Stanford T, Lee H, Fraysse F, Metcalf B, Mouatt B, Bennell K. The EPIPHA-KNEE trial: Explaining Pain to target unhelpful pain beliefs to Increase PHysical Activity in KNEE osteoarthritis - a protocol for a multicentre, randomised controlled trial with clinical- and cost-effectiveness analysis. BMC Musculoskelet Disord. 2021 Aug 28;22(1):738. doi: 10.1186/s12891-021-04561-6. PMID 34454458
- [Background] Rakel B, Cooper N, Adams HJ, Messer BR, Frey Law LA, Dannen DR, Miller CA, Polehna AC, Ruggle RC, Vance CG, Walsh DM, Sluka KA. A new transient sham TENS device allows for investigator blinding while delivering a true placebo treatment. J Pain. 2010 Mar;11(3):230-8. doi: 10.1016/j.jpain.2009.07.007. Epub 2009 Nov 27. PMID 19945354
- [Background] Mitchell UH, Stoneman P, Larson RE, Page GL. The Construction of Sham Dry Needles and Their Validity. Evid Based Complement Alternat Med. 2018 Jun 14;2018:9567061. doi: 10.1155/2018/9567061. eCollection 2018. PMID 30013605
- [Background] Fingleton C, Smart K, Moloney N, Fullen BM, Doody C. Pain sensitization in people with knee osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Jul;23(7):1043-56. doi: 10.1016/j.joca.2015.02.163. Epub 2015 Mar 5. PMID 25749012
- [Background] Shim JW, Jung JY, Kim SS. Effects of Electroacupuncture for Knee Osteoarthritis: A Systematic Review and Meta-Analysis. Evid Based Complement Alternat Med. 2016;2016:3485875. doi: 10.1155/2016/3485875. Epub 2016 Oct 13. PMID 27818699
- [Background] Dunning J, Butts R, Young I, Mourad F, Galante V, Bliton P, Tanner M, Fernandez-de-Las-Penas C. Periosteal Electrical Dry Needling as an Adjunct to Exercise and Manual Therapy for Knee Osteoarthritis: A Multicenter Randomized Clinical Trial. Clin J Pain. 2018 Dec;34(12):1149-1158. doi: 10.1097/AJP.0000000000000634. PMID 29864043
- [Background] Pisters MF, Veenhof C, van Meeteren NL, Ostelo RW, de Bakker DH, Schellevis FG, Dekker J. Long-term effectiveness of exercise therapy in patients with osteoarthritis of the hip or knee: a systematic review. Arthritis Rheum. 2007 Oct 15;57(7):1245-53. doi: 10.1002/art.23009. PMID 17907210
- [Background] Moseley GL, Butler DS. Fifteen Years of Explaining Pain: The Past, Present, and Future. J Pain. 2015 Sep;16(9):807-13. doi: 10.1016/j.jpain.2015.05.005. Epub 2015 Jun 5. PMID 26051220
- [Background] Kroon FP, van der Burg LR, Buchbinder R, Osborne RH, Johnston RV, Pitt V. Self-management education programmes for osteoarthritis. Cochrane Database Syst Rev. 2014 Jan 15;2014(1):CD008963. doi: 10.1002/14651858.CD008963.pub2. PMID 24425500
- [Background] Stanton TR, Karran EL, Butler DS, Hull MJ, Schwetlik SN, Braithwaite FA, Jones HG, Moseley GL, Hill CL, Tomkins-Lane C, Maher C, Bennell K. A pain science education and walking program to increase physical activity in people with symptomatic knee osteoarthritis: a feasibility study. Pain Rep. 2020 Sep 24;5(5):e830. doi: 10.1097/PR9.0000000000000830. eCollection 2020 Sep-Oct. PMID 33490835